CLINICAL TRIAL: NCT03697070
Title: INtelligent Stewardship Prompts to Improve Real-time Empiric Antibiotic Selection for Patients With Pneumonia
Brief Title: The INSPIRE-ASP PNA Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard Pilgrim Health Care (Other)
Collaborators: Hospital Corporation of America (Industry); University of California, Irvine (Other); University of Massachusetts, Amherst (Other); Brigham and Women's Hospital (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Richard Platt, Professor and Chair, Department of Population Medicine, Harvard Pilgrim Health Care
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PH000619B_PNA
Record Dates: First submitted 2018-10-03; First posted 2018-10-05 (Actual); Results first posted 2025-01-29 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2024-12

CONDITIONS: Pneumonia
Keywords: PNA; CPOE; Empiric Therapy
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: This cluster-randomized trial will assess a novel quality improvement antibiotic stewardship strategy for empiric antibiotic selection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care (Active Comparator): Continued routine antibiotic stewardship strategies.
  Interventions: Other: Routine Care
- INSPIRE CPOE Smart Prompt (Active Comparator): Use of a computerized physician order entry (CPOE) smart prompt alert to guide empiric choice of antibiotics for PNA in non-ICU patients in the first 3 days of hospitalization.
  Interventions: Other: INSPIRE CPOE Smart Prompt

INTERVENTIONS:
Other: INSPIRE CPOE Smart Prompt — Quality improvement intervention: computerized physician order entry (CPOE) decision support alert that provides physicians with patient-specific risk estimate of having PNA due to a multidrug resistant organism (MDRO) and recommends appropriate antibiotic choice for non-ICU patients in the first 3 days of hospitalization.
  Continuation of other antibiotic stewardship activities in accordance with national standards.
  Arms: INSPIRE CPOE Smart Prompt
Other: Routine Care — Routine Antibiotic Stewardship Arm - Continuation of all antibiotic stewardship activities in accordance with national standards.
  Arms: Routine Care

SUMMARY:
The INSPIRE-ASP PNA trial is a cluster-randomized controlled trial of HCA hospitals comparing routine empiric antibiotic stewardship practices with real-time precision medicine computerized physician order entry smart prompts providing the probability that a non-critically ill adult admitted with PNA is infected with a resistant pathogen.

Note: that enrolled "subjects" represents 59 individual HCA hospitals that have been randomized.

ELIGIBILITY:
Facility Inclusion Criteria:

* HCA hospitals admitting adults with PNA
* Facility use of MEDITECH as their electronic health record system

Facility Exclusion Criteria:

-

Note: unit of randomization is the hospital, however the CPOE alert intervention will calculate risk estimates for adults age >=18 admitted to non-ICU wards and who are ordered to receive extended-spectrum antibiotics for PNA. Prisoners were excluded from prompts and analysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44780 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2024-05-16 (Actual); Study Completion 2024-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shruti Gohil, MD, MPH, Study Director — UC Irvine Div Infectious Diseases; Susan Huang, MD, MPH, Principal Investigator — UC Irvine Div Infectious Diseases; Richard Platt, MD, MS, Principal Investigator — Harvard Pilgrim Health Care Institute
Locations (59):
- United States (59):
  - Riverside Community Hospital, Riverside, California
  - Regional Medical Center of San Jose, San Jose, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Swedish Medical Center, Denver, Colorado
  - Sky Ridge Medical Center, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Brandon Regional, Brandon, Florida
  - Fort Walton Medical Center, Fort Walton Beach, Florida
  - North Florida Regional Medical Center, Gainesville, Florida
  - Osceola Regional Medical Center, Kissimmee, Florida
  - Poinciana Medical Center, Kissimmee, Florida
  - Lake City Medical Center, Lake City, Florida
  - Largo Medical Center, Largo, Florida
  - Northwest Medical Center, Margate, Florida
  - Kendall Regional Medical Center, Miami, Florida
  - Twin Cities Hospital, Niceville, Florida
  - Putnam Community Medical Center, Palatka, Florida
  - Gulf Coast Medical Center, Panama City, Florida
  - Westside Regional Medical Center, Plantation, Florida
  - Fawcett Memorial Hospital, Port Charlotte, Florida
  - St. Lucie Medical Center, Port Saint Lucie, Florida
  - Central Florida Regional Hospital, Sanford, Florida
  - Doctor's Hospital Sarasota, Sarasota, Florida
  - Capital Regional Medical Center, Tallahassee, Florida
  - Medical Center of Trinity, Trinity, Florida
  - Cartersville Medical Center, Cartersville, Georgia
  - Fairview Park, Dublin, Georgia
  - Redmond Regional Medical Center, Rome, Georgia
  - West Valley Medical Center, Caldwell, Idaho
  - Terre Haute Regional Hospital, Terre Haute, Indiana
  - Tulane University Hospital & Clinic, New Orleans, Louisiana
  - Centerpoint Medical Center, Independence, Missouri
  - Research Medical Center, Kansas City, Missouri
  - Southern Hills Hospital - Vegas, Las Vegas, Nevada
  - TriStar Horizon Medical Center, Dickson, Tennessee
  - Stonecrest Medical Center, Nashville, Tennessee
  - South Austin Hospital, Austin, Texas
  - St. David's Medical Center, Austin, Texas
  - Valley Regional Medical Center, Brownsville, Texas
  - Conroe Regional Medical Center, Conroe, Texas
  - Corpus Christi Medical Center (Doctor's, Bay Area, and The Heart Hospital Campuses), Corpus Christi, Texas
  - Medical City Denton, Denton, Texas
  - Medical City Fort Worth, Fort Worth, Texas
  - West Houston Medical Center, Houston, Texas
  - Kingwood Medical Center, Kingwood, Texas
  - Rio Grande Regional Hospital, McAllen, Texas
  - North Hills Hospital, North Richland Hills, Texas
  - Bayshore Medical Center, Pasadena, Texas
  - Medical City Plano, Plano, Texas
  - Round Rock Hospital, Round Rock, Texas
  - Metropolitan Methodist Hospital, San Antonio, Texas
  - Clearlake Regional Medical Center, Webster, Texas
  - LewisGale Hospital - Montgomery, Blacksburg, Virginia
  - John Randolph Medical Center, Hopewell, Virginia
  - LewisGale Hospital - Pulaski, Pulaski, Virginia
  - Reston Hospital, Reston, Virginia
  - CJW Medical Center (Chippenham & Johnston Willis Campuses), Richmond, Virginia
  - Henrico Doctors' Hospital (Forest, Retreat, and Parham Campuses), Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gohil SK, Septimus E, Kleinman K, Varma N, Avery TR, Heim L, Rahm R, Cooper WS, Cooper M, McLean LE, Nickolay NG, Weinstein RA, Burgess LH, Coady MH, Rosen E, Sljivo S, Sands KE, Moody J, Vigeant J, Rashid S, Gilbert RF, Smith KN, Carver B, Poland RE, Hickok J, Sturdevant SG, Calderwood MS, Weiland A, Kubiak DW, Reddy S, Neuhauser MM, Srinivasan A, Jernigan JA, Hayden MK, Gowda A, Eibensteiner K, Wolf R, Perlin JB, Platt R, Huang SS. Stewardship Prompts to Improve Antibiotic Selection for Pneumonia: The INSPIRE Randomized Clinical Trial. JAMA. 2024 Jun 18;331(23):2007-2017. doi: 10.1001/jama.2024.6248. PMID 38639729

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 59 out of 143 HCA Healthcare hospitals were recruited for this trial. There was a 15 month intervention period from April 1, 2019 through June 30, 2020.
Pre-assignment Details: 44,780 patients were involved in the intervention period from the 59 participating hospitals.
Units Other Than Participants: Hospitals
Groups:
- Arm 1: Routine Stewardship: Continuation of all antibiotic stewardship activities in accordance with national standards.
- Arm 2: CPOE Bundle: Use of a computerized physician order entry (CPOE) smart prompt alert to guide empiric choice of antibiotics for PNA in non-ICU patients in the first 3 days of hospitalization.
Period: Overall Study
Arm/Group | Arm 1: Routine Stewardship | Arm 2: CPOE Bundle
Started | 21998; 30 Hospitals | 22782; 29 Hospitals
Completed | 21998; 30 Hospitals | 22782; 29 Hospitals
Not Completed | 0; 0 Hospitals | 0; 0 Hospitals

BASELINE CHARACTERISTICS:
Population: Number of participant totals reflect total intervention participants. 59 hospitals were randomized to a study group, 29 began the assigned intervention and 30 continued routine care.
Groups:
- Arm 2: CPOE Bundle: Use of a computerized physician order entry (CPOE) smart prompt alert to guide empiric choice of antibiotics for PNA in non-ICU patients in the first 3 days of hospitalization.
  INSPIRE CPOE Smart Prompt: Quality improvement intervention: computerized physician order entry (CPOE) decision support alert that provides physicians with patient-specific risk estimate of having PNA due to a multidrug resistant organism (MDRO) and recommends appropriate antibiotic choice for non-ICU patients in the first 3 days of hospitalization.
  Continuation of other antibiotic stewardship activities in accordance with national standards.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Routine Stewardship | Arm 2: CPOE Bundle | Total
Number analyzed (Participants) | 21998 | 22782 | 44780
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.4 (17.3) | 68.0 (17.0) | 68.0 (17.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Small differences in the number of patients with various characteristics reflect missing data in the electronic health record.
  Participants
    number analyzed (Participants) | 21945 | 22734 | 44679
    Female | 11400 | 11768 | 23168
    Male | 10545 | 10966 | 21511
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Small differences in the number of patients with various characteristics reflect missing data in the electronic health record.
  Participants
    Race: number analyzed (Participants) | 19161 | 21417 | 40578
    Race: Black | 2848 | 2908 | 5756
    Race: White | 15415 | 17205 | 32620
    Race: Other | 898 | 1304 | 2202

OUTCOME MEASURES:

1. Primary Outcome: Extended-Spectrum Days Of Antibacterial Therapy (ES-DOT) Per Empiric Day
Description: The number of different extended-spectrum antibacterials received by the patient each empiric day-of-therapy (outcome measure unit), averaged over the empiric days (the first 3 days of hospitalization), summed across all participants. Note that Days-of-Therapy unit is a standardized national measure for antibacterial use in hospitals. For clarity the calculation is as follows: we define a DOT for a particular ES antibiotic as a day in which any number of doses of that antibiotic is given. Different ES antibiotics are summed across the empiric days for each patient admission, then divided by the empiric days for that patient-admission to determine each admission's DOT per at-risk day. If an admission is less than 3 days, only the number of days the patient is admitted will contribute to the numerator and denominator.
Time Frame: First 3 days of hospitalization for each patient during 15-month intervention period
Population: The total number of participants analyzed reported here is from the intervention period.
Measure: Number; unit: Extended-Spectrum Days-of-Therapy
Arm/Group | Arm 1: Routine Stewardship | Arm 2: CPOE Bundle
Number analyzed (Participants) | 21998 | 22782
Extended-Spectrum Days-of-Therapy | 38690 | 27971

2. Secondary Outcome: Vancomycin Days of Antibacterial Therapy Per Empiric Day
Description: The number of days that Vancomycin is received by the patient averaged over the empiric days (the first 3 days of hospitalization), summed across all participants. Note that Days-of-Therapy unit is a standardized national measure for antibacterial use in hospitals. For clarity the calculation is as follows: we define a DOT for a particular ES antibiotic as a day in which any number of doses of that antibiotic is given. Different ES antibiotics are summed across the empiric days for each patient admission, then divided by the empiric days for that patient-admission to determine each admission's DOT per at-risk day. If an admission is less than 3 days, only the number of days the patient is admitted will contribute to the numerator and denominator.
Time Frame: First 3 days of hospitalization for each patient during 15-month intervention period
Population: The total number of participants analyzed reported here is from the intervention period.
Measure: Number; unit: Vancomycin Days-of-Therapy
Arm/Group | Arm 1: Routine Stewardship | Arm 2: CPOE Bundle
Number analyzed (Participants) | 21998 | 22782
Vancomycin Days-of-Therapy | 13778 | 10534

3. Secondary Outcome: Antipseudomonal Antibiotic Days Of Therapy (ES-DOT) Per Empiric Day
Description: The number of different antipseudomonals received by the patient each empiric day of therapy, averaged over the empiric days (the first 3 days of hospitalization), summed across all participants. Note that Days-of-Therapy unit is a standardized national measure for antibacterial use in hospitals. For clarity the calculation is as follows: we define a DOT for a particular ES antibiotic as a day in which any number of doses of that antibiotic is given. Different ES antibiotics are summed across the empiric days for each patient admission, then divided by the empiric days for that patient-admission to determine each admission's DOT per at-risk day. If an admission is less than 3 days, only the number of days the patient is admitted will contribute to the numerator and denominator.
Time Frame: First 3 days of hospitalization for each patient during 15-month intervention period
Population: The total number of participants analyzed reported here is from the intervention period.
Measure: Number; unit: Antipseudomonal Days-of-Therapy
Arm/Group | Arm 1: Routine Stewardship | Arm 2: CPOE Bundle
Number analyzed (Participants) | 21998 | 22782
Antipseudomonal Days-of-Therapy | 22683 | 15670

4. Other Pre Specified Outcome: Antibacterial Escalations [Safety Outcome 1]
Description: Days from start of standard-spectrum antibacterial until switch to extended-spectrum antibacterial during hospital stay, if that occurs. If it doesn't occur, the number of days is censored (capped) at the patient's hospital discharge or at the end of data collection. Almost all patients will be discharged before the end of trial data collection.
Time Frame: Duration of hospitalization for each patient during 15-month intervention period
Population: The mean number of days to event here is from the intervention period.
Measure: Mean (Standard Deviation); unit: Days to event
Arm/Group | Arm 1: Routine Stewardship | Arm 2: CPOE Bundle
Number analyzed (Participants) | 21998 | 22782
Days to event | 5.3 (3.8) | 6.1 (5.9)

5. Other Pre Specified Outcome: ICU Transfers [Safety Outcome 2]
Description: Days from hospital admission until transfer to ICU, if that occurs. If it doesn't occur, the number of days is censored (capped) at the patient's hospital discharge or at the end of data collection. Almost all patients will be discharged before the end of trial data collection.
Time Frame: Duration of hospitalization for each patient during 15-month intervention period
Population: The mean number of days to event here is from the intervention period.
Measure: Mean (Standard Deviation); unit: Days to event
Arm/Group | Arm 1: Routine Stewardship | Arm 2: CPOE Bundle
Number analyzed (Participants) | 21998 | 22782
Days to event | 6.5 (5.2) | 7.1 (5.9)

6. Other Pre Specified Outcome: Length-of-stay [Safety Outcome 3]
Description: Days from hospital admission until discharge. If the patient remains in the hospital at the end of the trial data collection, the number of days is censored (capped) at that time. Almost all patients will be discharged before the end of trial data collection.
Time Frame: Duration of hospitalization for each patient during 15-month intervention period
Population: The mean number of days to event here is from the intervention period.
Measure: Mean (Standard Deviation); unit: Days to event
Arm/Group | Arm 1: Routine Stewardship | Arm 2: CPOE Bundle
Number analyzed (Participants) | 21998 | 22782
Days to event | 6.8 (5.9) | 7.1 (6.9)

7. Other Pre Specified Outcome: Extended-Spectrum Days of Therapy With Inpatient Extended-Spectrum (ES) Antibacterial Treatment After Empiric Period
Description: The summed number of different ES antibacterials received each day, measured repeatedly on or after 4 calendar days of admission and divided by the number of days from hospital day 4 through discharge.
  Note: this outcome is intended for a secondary manuscript.
Time Frame: 15 month intervention
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Empiric and Total Antibacterial Costs
Description: Empiric and total antibacterial costs during hospitalization.
  Note: this outcome is intended for a secondary manuscript.
Time Frame: 15 month intervention
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Incidence of Hospital-Onset C. Difficile
Description: Hospital-onset C. difficile positive tests (specimen obtained) after 3 calendar days of admission during hospitalization.
  Note: this outcome is intended for a secondary manuscript.
Time Frame: 15 month intervention
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Incidence of Hospital-Onset MDRO-Positive Cultures
Description: Newly-detected hospital-onset MDRO-positive cultures (on or after 3 calendar days of admission). Includes total MDRO and specific MDRO subsets.
  Note: this outcome is intended for a secondary manuscript.
Time Frame: 15 month intervention
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Fluoroquinolone (FQ) Days of Therapy Per Empiric and Total At-risk Days
Description: The summed number of different fluoroquinolone antibacterials received each day, measured repeatedly over (1) the first three days (empiric) of an admission and divided by the number of days of the admission and (2) all days of an admission divided by the total number of admission days.
  Note: this outcome is intended for a secondary manuscript.
Time Frame: 15 month intervention
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 15 Months
Arm/Group | Arm 1: Routine Stewardship | Arm 2: CPOE Bundle
All-Cause Mortality (participants affected / at risk) | 0/21998 | 0/22782
Serious Adverse Events (participants affected / at risk) | 0/21998 | 0/22782
Other Adverse Events (participants affected / at risk) | 0/21998 | 0/22782

LIMITATIONS AND CAVEATS:
[Not Specified]

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT03697070/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT03697070/SAP_001.pdf